CLINICAL TRIAL: NCT05482724
Title: Treatment of Emotional Disorders in Spanish Children: Efficacy of Super Skills for Life Transdiagnostic Treatment
Brief Title: Super Skills for Life Effectiveness in Clinical Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Mireia Orgilés Amorós, Director, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/034
Record Dates: First submitted 2022-07-22; First posted 2022-08-01 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Depressive Disorder; Depressive Symptoms; Trauma and Stressor Related Disorders; Anxiety Disorders and Symptoms; Anxiety Disorders; Mood Disorders; Emotional Disorder
MeSH Terms: conditions — Depressive Disorder; Depression; Trauma and Stressor Related Disorders; Anxiety Disorders; Mood Disorders

STUDY DESIGN:
Intervention Model Description: Participants who met the inclusion criteria and underwent thorough the baseline assessment were randomly allocated to the conditions of the intervention group and the wait-list control group. Participants in the wait-list group (WLC) received no phycological (public or private) intervention during the eight-week duration of the program. Children and parents in both groups would complete the same series of measures at about the same time (pre-test and after eight weeks). Children in WLC group will receive the intervention once the follow-up visit is completed.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Super Skills for Life intervention group
  Interventions: Behavioral: Super Skills for Life
- Wait-list group (No Intervention): Group without any intervention. Participants in the wait-list group received no phycological (public or private) intervention during the eight-week duration of the SSL program. They were informed that children in this group will receive the intervention once the follow-up visit is completed.

INTERVENTIONS:
Behavioral: Super Skills for Life — Structured and manualized intervention with a manual for the therapist and a workbook for the children.
  Spanish version of Super Skills for Life group program: Orgilés, M., Espada, J.P., Ollendick, T.H. & Essau, C. (2022). Programa Super Skills. Manual del aplicador. Elche, ES: Universidad Miguel Hernández.
  The intervention was administered by a trained clinical psychologist in SSL. Sessions were held after school hours once a week for eight weeks, with each session lasting approximately one hour. The contents of the program were covered through playful activities in groups of 4 to 6 children
  Arms: Intervention group

SUMMARY:
Super Skills for Life (SSL) is a transdiagnostic cognitive-behavioral protocol developed for children aged 6 to 12 with anxiety and comorbid problems (e.g., depression, low self-esteem, and lack of social skills).

SSL consists of eight sessions targeting common risk factors for internalizing disorders such as cognitive distortions, avoidance, emotional management, low self-esteem, social skills deficits and coping strategies.

The aim of the study is to investigate the short- and long-term effects of SSL on internalizing and externalizing symptoms in Spanish children attending the Child and Adolescent Mental Health Services.

DETAILED DESCRIPTION:
To validate eligibility children and their parents will complete several psychometrically robust and developmentally appropriate measures. Participants meeting inclusion criteria will be randomly allocated to the conditions of the intervention group and the wait-list control group.

Parents and children from both groups will complete the same measures at baseline and post-treatment.

Parents and children from SSL will also complete these measures at 3 months follow-up, 6 months follow-up and 12 months follow-up.

The investigators will assess the benefits from pre-test to post-test in children participating in SSL compared to those in a wait-list control group on DSM-5 diagnostic remission, anxiety symptoms, anxiety impairment, depressive symptoms, self-esteem, behavioral problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior.

The investigators will also assess these variables in the intervention group at 3 months, 6 months, and 12 months follow-up.

Ultimately, the goal of the study is to explore whether SSL can be a cost-effective psychological intervention for emotional disorders in the Spanish National Health System.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 - 12.
* Primary diagnosis of an anxiety disorder, a depressive disorder, and/or trauma- or stress-related disorder with anxiety and/or depressive symptoms.
* Speaking, reading, writing and understanding Spanish.
* Caregivers agree to attend all sessions and to receive feedback and suggestions.

Exclusion Criteria:

* Intellectual disability, behavioral symptoms, or autism spectrum symptoms whose severity precluded continued treatment.
* The child is at the same time in psychological treatment.
* The child is not on a stable dose of medication for at least 1 month prior to baseline assessment.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline diagnosis based on DSM-5 criteria to immediately after the intervention | baseline and immediately after the intervention
  Measured by Schedule for affective disorders and schizophrenia for schoolage youths-present and lifetime version (K-SADS-PL). The K-SADS-PL is a semi-structured interview for children and adolescents aged 6 to 18 years according to DSM-IV criteria. Additional questions were included in this study to obtain a diagnosis according to the current DSM-5 classification.
Diagnosis based on DSM-5 criteria at 3 months | 3 months after the intervention
  Measured by Schedule for affective disorders and schizophrenia for schoolage youths-present and lifetime version (K-SADS-PL). The K-SADS-PL is a semi-structured interview for children and adolescents aged 6 to 18 years according to DSM-IV criteria. Additional questions were included in this study to obtain a diagnosis according to the current DSM-5 classification.
Diagnosis based on DSM-5 criteria at 6 months | 6 months after the intervention
  Measured by Schedule for affective disorders and schizophrenia for schoolage youths-present and lifetime version (K-SADS-PL). The K-SADS-PL is a semi-structured interview for children and adolescents aged 6 to 18 years according to DSM-IV criteria. Additional questions were included in this study to obtain a diagnosis according to the current DSM-5 classification.
Diagnosis based on DSM-5 criteria at 1 year | 1 year after the intervention
  Measured by Schedule for affective disorders and schizophrenia for schoolage youths-present and lifetime version (K-SADS-PL). The K-SADS-PL is a semi-structured interview for children and adolescents aged 6 to 18 years according to DSM-IV criteria. Additional questions were included in this study to obtain a diagnosis according to the current DSM-5 classification.
Change from baseline depression symptoms to immediately after the intervention | baseline and immediately after the intervention
  Measured by Child Depression Inventory (CDI). It assess depressive symptoms experienced in the past two weeks. The CDI provides an overall score (minimum value 0, maximum value 54) and two dimensions values: dysphoria (minimum value 0, maximum value 34), and negative self-esteem (minimum value 0, maximum value 20). Higher scores indicate more severe symptoms.
Depression symptoms at 3 months | 3 months after the intervention
  Measured by Child Depression Inventory (CDI). It assess depressive symptoms experienced in the past two weeks. The CDI provides an overall score (minimum value 0, maximum value 54) and two dimensions values: dysphoria (minimum value 0, maximum value 34), and negative self-esteem (minimum value 0, maximum value 20). Higher scores indicate more severe symptoms.
Depression symptoms at 6 months | 6 months after the intervention
  Measured by Child Depression Inventory (CDI). It assess depressive symptoms experienced in the past two weeks. The CDI provides an overall score (minimum value 0, maximum value 54) and two dimensions values: dysphoria (minimum value 0, maximum value 34), and negative self-esteem (minimum value 0, maximum value 20). Higher scores indicate more severe symptoms.
Depression symptoms at 1 year | 1 year after the intervention
  Measured by Child Depression Inventory (CDI). It assess depressive symptoms experienced in the past two weeks. The CDI provides an overall score (minimum value 0, maximum value 54) and two dimensions values: dysphoria (minimum value 0, maximum value 34), and negative self-esteem (minimum value 0, maximum value 20). Higher scores indicate more severe symptoms.
Change from baseline parent-reported anxiety symptoms to immediately after the intervention | baseline and immediately after the intervention
  Measured by Spence Children's Anxiety Scale Parent Report (SCAS-P). SCAS-P measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety and specific fears). Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 114. Higher scores indicating greater severity of symptoms.
Change from baseline children's reported anxiety symptoms to immediately after the intervention | baseline and immediately after the intervention
  Measured by Spence Children's Anxiety Scale Child Report (SCAS). SCAS measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety and specific fears). Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 114. Higher scores indicating greater severity of symptoms.
Parent-reported anxiety symptoms at 3 months | 3 months after the intervention
  Measured by Spence Children's Anxiety Scale Parent Report (SCAS-P). SCAS-P measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety and specific fears). Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 114. Higher scores indicating greater severity of symptoms.
Children's reported anxiety symptoms at 3 months | 3 months after the intervention
  Measured by Spence Children's Anxiety Scale Child Report (SCAS). SCAS measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety and specific fears). Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 114. Higher scores indicating greater severity of symptoms.
Parent-reported anxiety symptoms at 6 months | 6 months after the intervention
  Measured by Spence Children's Anxiety Scale Parent Report (SCAS-P). SCAS-P measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety and specific fears). Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 114. Higher scores indicating greater severity of symptoms.
Children's reported anxiety symptoms at 6 months | 6 months after the intervention
  Measured by Spence Children's Anxiety Scale Child Report (SCAS). SCAS measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety and specific fears). Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 114. Higher scores indicating greater severity of symptoms.
Parent-reported anxiety symptoms at 1 year | 1 year after the intervention
  Measured by Spence Children's Anxiety Scale Parent Report (SCAS-P). SCAS-P measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety and specific fears). Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 114. Higher scores indicating greater severity of symptoms.
Children's reported anxiety symptoms at 1 year | 1 year after the intervention
  Measured by Spence Children's Anxiety Scale Child Report (SCAS). SCAS measures symptoms severity of the DSM-IV anxiety disorders in children (subscales: total, panic and agoraphobia, generalized anxiety disorder, obsessive-compulsive disorder, social phobia, separation anxiety and specific fears). Symptom frequency is recorded on a 3-point Likert scale from 0 (never) to 3 (always). This yields a minimum possible score of 0 and a maximum possible score of 114. Higher scores indicating greater severity of symptoms.
Change from baseline parent-reported anxiety-related interference to immediately after the intervention | baseline and immediately after the intervention
  Measured by Child Anxiety Life Interference Scale Parent Report (CALIS-P). It assesses life interference and impairment related to anxiety in the child's school, social, and home/family settings. Scores range from a minimum value of 0 to a maximun value of 64. Higher scores indicate larger child anxiety-related interference.
Change from baseline children's reported anxiety-related interference to immediately after the intervention | baseline and immediately after the intervention
  Measured by Child Anxiety Life Interference Scale Child Report (CALIS-C). It assesses life interference and impairment related to anxiety in the child's school, social, and home/family settings. Scores range from a minimum value of 0 to a maximun value of 36. Higher scores indicate larger child anxiety-related interference.
Parent-reported anxiety-related interference at 3 months | 3 months after the intervention
  Measured by Child Anxiety Life Interference Scale Parent Report (CALIS-P). It assesses life interference and impairment related to anxiety in the child's school, social, and home/family settings. Scores range from a minimum value of 0 to a maximun value of 64. Higher scores indicate larger child anxiety-related interference.
Children's reported anxiety-related interference at 3 months | 3 months after the intervention
  Measured by Child Anxiety Life Interference Scale Child Report (CALIS-C). It assesses life interference and impairment related to anxiety in the child's school, social, and home/family settings. Scores range from a minimum value of 0 to a maximun value of 36. Higher scores indicate larger child anxiety-related interference.
Parent-reported anxiety-related interference at 6 months | 6 months after the intervention
  Measured by Child Anxiety Life Interference Scale Parent Report (CALIS-P). It assesses life interference and impairment related to anxiety in the child's school, social, and home/family settings. Scores range from a minimum value of 0 to a maximun value of 64. Higher scores indicate larger child anxiety-related interference.
Children's reported anxiety-related interference at 6 months | 6 months after the intervention
  Measured by Child Anxiety Life Interference Scale Child Report (CALIS-C). It assesses life interference and impairment related to anxiety in the child's school, social, and home/family settings. Scores range from a minimum value of 0 to a maximun value of 36. Higher scores indicate larger child anxiety-related interference.
Parent-reported anxiety-related interference at 1 year | 1 year after the intervention
  Measured by Child Anxiety Life Interference Scale Parent Report (CALIS-P). It assesses life interference and impairment related to anxiety in the child's school, social, and home/family settings. Scores range from a minimum value of 0 to a maximun value of 64. Higher scores indicate larger child anxiety-related interference.
Children's reported anxiety-related interference at 1 year | 1 year after the intervention
  Measured by Child Anxiety Life Interference Scale Child Report (CALIS-C). It assesses life interference and impairment related to anxiety in the child's school, social, and home/family settings. Scores range from a minimum value of 0 to a maximun value of 36. Higher scores indicate larger child anxiety-related interference.

SECONDARY OUTCOMES:
Change from baseline children's reported global mental health symptoms to immediately after the intervention | baseline and immediately after the intervention
  Measured by Strengths and Difficulties Questionnaire Child Report (SDQ). It was designed to measure children's overall difficulties (minimum value 0 and maximum value 40) and positive attributes across five subscales (minimum value 0 and maximun value 10): Emotional symptoms (e.g., anxiety and depression), Conduct problems, Hyperactivity/Inattention, Peer relationships (difficulties), and Pro-social behavior. . Higher scores indicate higher levels of difficulties, except on the prosocial subscale, where higher scores reflect a more positive attribute.
Change from baseline parent's reported global mental health symptoms to immediately after the intervention | baseline and immediately after the intervention
  Measured by Strengths and Difficulties Questionnaire Parent Report (SDQ-P). It was designed to measure children's overall difficulties (minimum value 0 and maximum value 40) and positive attributes across five subscales (minimum value 0 and maximum value 10): Emotional symptoms (e.g., anxiety and depression), Conduct problems, Hyperactivity/Inattention, Peer relationships (difficulties), and Pro-social behavior. . Higher scores indicate higher levels of difficulties, except on the prosocial subscale, where higher scores reflect a more positive attribute.
Children's reported global mental health symptoms at 3 months | 3 months after the intervention
  Measured by Strengths and Difficulties Questionnaire Child Report (SDQ). It was designed to measure children's overall difficulties (minimum value 0 and maximum value 40) and positive attributes across five subscales (minimum value 0 and maximun value 10): Emotional symptoms (e.g., anxiety and depression), Conduct problems, Hyperactivity/Inattention, Peer relationships (difficulties), and Pro-social behavior. . Higher scores indicate higher levels of difficulties, except on the prosocial subscale, where higher scores reflect a more positive attribute.
Parent's reported global mental health symptoms at 3 months | 3 months after the intervention
  Measured by Strengths and Difficulties Questionnaire Parent Report (SDQ-P). It was designed to measure children's overall difficulties (minimum value 0 and maximum value 40) and positive attributes across five subscales (minimum value 0 and maximum value 10): Emotional symptoms (e.g., anxiety and depression), Conduct problems, Hyperactivity/Inattention, Peer relationships (difficulties), and Pro-social behavior. . Higher scores indicate higher levels of difficulties, except on the prosocial subscale, where higher scores reflect a more positive attribute.
Children's reported global mental health symptoms at 6 months | 6 months after the intervention
  Measured by Strengths and Difficulties Questionnaire Child Report (SDQ). It was designed to measure children's overall difficulties (minimum value 0 and maximum value 40) and positive attributes across five subscales (minimum value 0 and maximun value 10): Emotional symptoms (e.g., anxiety and depression), Conduct problems, Hyperactivity/Inattention, Peer relationships (difficulties), and Pro-social behavior. . Higher scores indicate higher levels of difficulties, except on the prosocial subscale, where higher scores reflect a more positive attribute.
Parent's reported global mental health symptoms at 6 months | 6 months after the intervention
  Measured by Strengths and Difficulties Questionnaire Parent Report (SDQ-P). It was designed to measure children's overall difficulties (minimum value 0 and maximum value 40) and positive attributes across five subscales (minimum value 0 and maximum value 10): Emotional symptoms (e.g., anxiety and depression), Conduct problems, Hyperactivity/Inattention, Peer relationships (difficulties), and Pro-social behavior. . Higher scores indicate higher levels of difficulties, except on the prosocial subscale, where higher scores reflect a more positive attribute.
Children's reported global mental health symptoms at 1 year | 1 year after the intervention
  Measured by Strengths and Difficulties Questionnaire Child Report (SDQ). It was designed to measure children's overall difficulties (minimum value 0 and maximum value 40) and positive attributes across five subscales (minimum value 0 and maximun value 10): Emotional symptoms (e.g., anxiety and depression), Conduct problems, Hyperactivity/Inattention, Peer relationships (difficulties), and Pro-social behavior. . Higher scores indicate higher levels of difficulties, except on the prosocial subscale, where higher scores reflect a more positive attribute.
Parent's reported global mental health symptoms at 1 year | 1 year after the intervention
  Measured by Strengths and Difficulties Questionnaire Parent Report (SDQ-P). It was designed to measure children's overall difficulties (minimum value 0 and maximum value 40) and positive attributes across five subscales (minimum value 0 and maximum value 10): Emotional symptoms (e.g., anxiety and depression), Conduct problems, Hyperactivity/Inattention, Peer relationships (difficulties), and Pro-social behavior. . Higher scores indicate higher levels of difficulties, except on the prosocial subscale, where higher scores reflect a more positive attribute.
Change from baseline self-esteem to immediately after the intervention | baseline and immediately after the intervention
  Self-Concept Form 5 (AF-5). It measures global satisfaction with self-concept (minimum value 0 and maximum value 120) and five dimensions (minimum value 0 and maximum value 24): Social (performance in social relationships); Academic/Professional (student/worker role); Emotional (perception of emotional state in general and in specific situations); Family (participation and integration into the family unit); and Physical self-concept (appearance and physical condition). Higher scores indicate greater satisfaction with self-image.
Self-esteem at 3 months | 3 months after the intervention
  Self-Concept Form 5 (AF-5). It measures global satisfaction with self-concept (minimum value 0 and maximum value 120) and five dimensions (minimum value 0 and maximum value 24): Social (performance in social relationships); Academic/Professional (student/worker role); Emotional (perception of emotional state in general and in specific situations); Family (participation and integration into the family unit); and Physical self-concept (appearance and physical condition). Higher scores indicate greater satisfaction with self-image.
Self-esteem at 6 months | 6 months after the intervention
  Self-Concept Form 5 (AF-5). It measures global satisfaction with self-concept (minimum value 0 and maximum value 120) and five dimensions (minimum value 0 and maximum value 24): Social (performance in social relationships); Academic/Professional (student/worker role); Emotional (perception of emotional state in general and in specific situations); Family (participation and integration into the family unit); and Physical self-concept (appearance and physical condition). Higher scores indicate greater satisfaction with self-image.
Self-esteem at 1 year | 1 year after the intervention
  Self-Concept Form 5 (AF-5). It measures global satisfaction with self-concept (minimum value 0 and maximum value 120) and five dimensions (minimum value 0 and maximum value 24): Social (performance in social relationships); Academic/Professional (student/worker role); Emotional (perception of emotional state in general and in specific situations); Family (participation and integration into the family unit); and Physical self-concept (appearance and physical condition). Higher scores indicate greater satisfaction with self-image.
Perfectionism | pre-intervention
  Frost Multidimensional Perfectionism Scale (FMPS). A self-report measure with four sub-scales of perfectionism: concern over mistakes and doubts about actions, excessive concern with parents' expectations and evaluation, excessively high personal standards, concern with precision, order and organisation.
Changes from baseline health-related quality of life to immediately after the intervention | baseline and immediately after the intervention
  Health-Related Quality of Life Questionnaire for Children and Adolescents aged from 8 to 18 years (KIDSCREEN). It assess children's and parents' subjective health and well-being in 10 areas.
Health-related quality of life at 3 months | 3 months after the intervention
  Health-Related Quality of Life Questionnaire for Children and Adolescents aged from 8 to 18 years (KIDSCREEN). It assess children's and parents' subjective health and well-being in 10 areas.
Health-related quality of life at 6 months | 6 months after the intervention
  Health-Related Quality of Life Questionnaire for Children and Adolescents aged from 8 to 18 years (KIDSCREEN). It assess children's and parents' subjective health and well-being in 10 areas.
Health-related quality of life at 1 year | 1 year after the intervention
  Health-Related Quality of Life Questionnaire for Children and Adolescents aged from 8 to 18 years (KIDSCREEN). It assess children's and parents' subjective health and well-being in 10 areas.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Diego, Principal Investigator — Universidad Miguel Hernandez de Elche; Mireia Orgiles, Study Director — Universidad Miguel Hernandez de Elche
Locations (1):
- Hospital Clínico Universitario Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD
Supporting Information: SAP, Analytic Code
Time Frame: Starting after finishing all analysis and publication.
Access Criteria: Upon request and verification by the principal investigator to consult the available data. The use of the data for distribution in any format is not permitted.

REFERENCES:
- [Background] Essau CA, Olaya B, Sasagawa S, Pithia J, Bray D, Ollendick TH. Integrating video-feedback and cognitive preparation, social skills training and behavioural activation in a cognitive behavioural therapy in the treatment of childhood anxiety. J Affect Disord. 2014;167:261-7. doi: 10.1016/j.jad.2014.05.056. Epub 2014 Jun 4. PMID 24999861
- [Background] Essau CA, Sasagawa S, Jones G, Fernandes B, Ollendick TH. Evaluating the real-world effectiveness of a cognitive behavior therapy-based transdiagnostic program for emotional problems in children in a regular school setting. J Affect Disord. 2019 Jun 15;253:357-365. doi: 10.1016/j.jad.2019.04.036. Epub 2019 Apr 16. PMID 31078836
- [Background] Orgiles M, Fernandez-Martinez I, Espada JP, Morales A. Spanish version of Super Skills for Life: short- and long-term impact of a transdiagnostic prevention protocol targeting childhood anxiety and depression. Anxiety Stress Coping. 2019 Nov;32(6):694-710. doi: 10.1080/10615806.2019.1645836. Epub 2019 Jul 23. PMID 31334667
- [Background] Fernandez-Martinez I, Orgiles M, Morales A, Espada JP, Essau CA. One-Year follow-up effects of a cognitive behavior therapy-based transdiagnostic program for emotional problems in young children: A school-based cluster-randomized controlled trial. J Affect Disord. 2020 Feb 1;262:258-266. doi: 10.1016/j.jad.2019.11.002. Epub 2019 Nov 4. PMID 31733917
- [Background] Fernandez-Martinez I, Morales A, Espada JP, Orgiles M. Effects of Super Skills for Life on the social skills of anxious children through video analysis. Psicothema. 2020 May;32(2):229-236. doi: 10.7334/psicothema2019.240. PMID 32249749
- [Background] Melero S, Orgiles M, Espada JP, Morales A. Spanish version of Super Skills for Life in individual modality: Improvement of children's emotional well-being from a transdiagnostic approach. J Clin Psychol. 2021 Oct;77(10):2187-2202. doi: 10.1002/jclp.23148. Epub 2021 Apr 21. PMID 33882156
- [Background] Melero S, Morales A, Espada JP, Mendez X, Orgiles M. Effectiveness of Group vs. Individual Therapy to Decrease Peer Problems and Increase Prosociality in Children. Int J Environ Res Public Health. 2021 Apr 9;18(8):3950. doi: 10.3390/ijerph18083950. PMID 33918640
- [Background] Melero S, Morales A, Espada JP, Orgiles M. Improving Social Performance Through Video-feedback with Cognitive Preparation in Children with Emotional Problems. Behav Modif. 2022 Jul;46(4):755-781. doi: 10.1177/0145445521991098. Epub 2021 Jan 29. PMID 33511861
- [Background] Escribano S, Espada JP, Orgiles M, Morales A. Implementation fidelity for promoting the effectiveness of an adolescent sexual health program. Eval Program Plann. 2016 Dec;59:81-87. doi: 10.1016/j.evalprogplan.2016.08.008. Epub 2016 Aug 31. PMID 27614301
- [Background] Orgiles M, Melero S, Fernandez-Martinez I, Espada JP, Morales A. Effectiveness of Video-Feedback with Cognitive Preparation in Improving Social Performance and Anxiety through Super Skills for Life Programme Implemented in a School Setting. Int J Environ Res Public Health. 2020 Apr 18;17(8):2805. doi: 10.3390/ijerph17082805. PMID 32325756
- See also: University of Roehampton research for Super Skills for Life programme — https://www.superskillsforlife.com/